CLINICAL TRIAL: NCT05630560
Title: Common Factors, Responsiveness and Outcome in Psychotherapy (CROP): Study Protocol for an Observational Study of Psychotherapy in Private Practice
Brief Title: Common Factors, Responsiveness and Outcome in Psychotherapy
Acronym: CROP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Common Factors, Responsiveness and Outcome of Psychotherapy Study (Other)
Collaborators: University of Copenhagen (Other); The Health Foundation (Other); TRYG Foundation (Other); the Danish Psychological Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16-B-0269
Record Dates: First submitted 2022-11-11; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Mental Health; Psychological Distress; General Psychotherapy
Keywords: psychotherapy research; psychotherapy effect; psychotherapy process and outcome; therapist effects; therapy predictors and moderators; therapist responsiveness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychologists in Danish private practice: All psychologists with a Danish university degree in psychology who have registered themselves as seeing clients in private practice (app. 1,750) have been invited to participate in the study. Thus, the sample of psychologists consists of psychologists employed in the Danish practice sector, where clients obtain a refund of 60% of the psychologist's salary, as well as psychologists working privately without any reimbursement of their salaries. Each psychologist enrolled in the study has agreed to aim to recruit no less than 10 clients each for the study. We aim to include 100 psychologists, which will yield a sample of 1,000 clients beginning therapy.
  Interventions: Other: Psychotherapy treatment

INTERVENTIONS:
Other: Psychotherapy treatment — The psychotherapist will conduct psychotherapy as normally done by them in their practice. The treatment will thus be un-manualized and consist of a broad range of therapeutic orientations and treatment lengths.

SUMMARY:
The "Common Factors, Responsiveness and Outcome of Psychotherapy" (CROP) study is a naturalistic observational study at the University of Copenhagen (UCPH) carried out in cooperation with psychologists in the Danish practice sector or in private practice. The study aims to examine the contribution of client, therapist and treatment characteristics, as well as the role of therapists' responsiveness, on the process and outcome of psychotherapy. Participating psychologists and clients fill out background questionnaires prior to initiating therapy, and process data for each course of treatment is collected weekly and after each session while outcome data is collected at end of treatment and at three months follow-up. The psychologists are reimbursed DKK 1,000 per client that contributes to the study with at least three session questionnaires, which corresponds to the hourly salary of a psychologist in Danish private practice. All data is collected through an automated, online database to ensure appropriate anonymization and data management, and all participants give informed consent prior to participation. The CROP study has been approved by the UCPH's Department of Psychology's ethical review board and the Danish Data Protection Agency.

DETAILED DESCRIPTION:
The aim of the Common factors, Responsiveness and Outcome in Psychotherapy study (CROP) is to determine client and psychologist characteristics and therapeutic processes associated with the outcome of psychotherapy delivered by psychologists in the Danish practice sector or in private practice. The study addresses two main questions. First, how are specific characteristics of clients and psychologists related to the outcome of therapy and do these characteristics moderate the outcome of different psychotherapeutic approaches? Second, to what extent do therapists adapt their approach to client characteristics and preferences and how does such responsiveness impact the process and outcome of therapy? The results from the study are directly relevant to psychologists and will be disseminated nationwide during and after the end of the study.

The study is a naturalistic, observational study carried out in collaboration with psychologists in the Danish practice sector or in private practice. Self-report data is collected on the participating psychologists and their participating clients before psychotherapy, during psychotherapy (weekly and post-session) and after psychotherapy (at end of treatment and three months follow-up). The data is analyzed using multilevel modeling and structural equation modeling approaches.

The study design and data management procedure have been approved by the Research Ethics Board of the Department of Psychology, University of Copenhagen, and the Danish Data Protection Agency. All data are fully anonymized and stored in agreement with the Danish Act on Processing of Personal Data. All parts of the study are based on the principles of informed consent and clients are informed that they can terminate their participation in the study at any time without consequences to their treatment. The findings of the study will be presented in articles in international, peer-reviewed journals as well as to psychotherapy practitioners across Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 of age and in individual psychotherapy

Exclusion Criteria:

* severe psychoticism or other severe mental health issues.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, other
Study Population: All clients in individual psychotherapy aged 18 or older are eligible for the study, meaning that in principle all client diagnoses and referral reasons may be represented in the sample. However, in Denmark, reimbursement for psychological treatment in the practice sector is only provided for clients referred by their general practitioner for one of the 11 referral reasons and diagnoses presented below. Thus, clients meeting these characteristics are likely to be overrepresented within the sample.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in psychological symptoms measured by the BSI | Change in psychological symptoms from baseline until end-of-treatment (an average of 7 months).
  The Brief Symptom Inventory (BSI) is a self-report scale consisting of 53 items covering nine symptom dimensions: Somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.

SECONDARY OUTCOMES:
Change in symptoms measured by the Symptom Checklist-11 | Every week while the client is in therapy, up until 25 weeks of therapy.
  Symptom Checklist-11 (SCL-11) is a short, multidimensional outcome measure for the evaluation of therapeutic progress in psychotherapy, consisting of 11 items selected from the BSI using a stepwise item selection procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No participant data is planned to be shared with other researchers besides the CROP research team members.

REFERENCES:
- [Derived] Jacobsen CF, Igra L, Lunn S, Karstoft KI, Nielsen J, Lauritzen L, Falkenstrom F, Poulsen S. The association between therapist internal relational models, professional self-doubt, and coping strategies and the process and outcome of psychotherapy. Psychother Res. 2025 May 27:1-16. doi: 10.1080/10503307.2025.2506650. Online ahead of print. PMID 40424535
- [Derived] Jacobsen CF, Falkenstrom F, Karstoft KI, Igra L, Lunn S, Nielsen J, Lauritzen L, Poulsen S. Exploring the matching effect: The association between preference accommodation, the working alliance, and outcome in psychotherapy. J Consult Clin Psychol. 2025 Jun;93(6):443-456. doi: 10.1037/ccp0000955. PMID 40388150
- [Derived] Jacobsen CF, Falkenstrom F, Castonguay L, Nielsen J, Lunn S, Lauritzen L, Poulsen S. The relationship between attachment needs, earned secure therapeutic attachment and outcome in adult psychotherapy. J Consult Clin Psychol. 2024 Jul;92(7):410-421. doi: 10.1037/ccp0000900. PMID 39190445
- [Derived] Faye Jacobsen C, Karstoft KI, Falkenstrom F, Nielsen J, Lunn S, Poulsen S. Client preferences, therapy activities and preference-activity match as predictors of therapy outcome. Psychother Res. 2025 Jun;35(5):777-792. doi: 10.1080/10503307.2024.2353358. Epub 2024 May 21. PMID 38771973
- [Derived] Lauritzen LR, Faye Jacobsen C, Nielsen J, Lunn S, Mathiesen BB, Falkenstrom F, Poulsen S. Common factors, Responsiveness and Outcome in Psychotherapy (CROP): study protocol for a naturalistic prospective cohort study of psychotherapy in Denmark. BMJ Open. 2023 Jun 2;13(6):e072277. doi: 10.1136/bmjopen-2023-072277. PMID 37270190